CLINICAL TRIAL: NCT03544177
Title: Effects of Low-intensity Interval Walking With Blood Flow Restriction on Gait Speed and Functional Impairments in Patients With Severe Multiple Sclerosis: a Pilot Study
Brief Title: Effects of Low-intensity Interval Walking With Blood Flow Restriction on Functional Capacity in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170783
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
Keywords: mobility; exercise therapy; blood flow restricted exercise; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Single-center pilot randomized parallel group clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcome measures assessors, blinded to group allocation, will not have access to the randomization list and unblinding will not be possible for these researchers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFR-Walking (Experimental): Interval walking training with blood flow restriction.
  Interventions: Other: BFR-Walking
- Conventional therapy (Active Comparator): Conventional therapy
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: BFR-Walking — Participants will perform 12 training sessions over 6 weeks, including a 10-minute warm up and cool down period. Patients will perform 5 six-minute bouts of over ground intermittent walking exercise (1-minute walk/rest) with their habitual walking device at a prescribed speed maintained by a metronome, starting from 60 steps/minute. A fixed resting period of 3 minutes will follow each walking bout. During walking, participants will wear BFR bands at both tights. Before every walking bout, the bands will be tightened at a low intensity (max 40% of blood systolic pressure) and untied at the end of every walking bout when patients will be asked to grade their RPE (Borg Scale). Walking speed will be weekly increased by 3 steps/minute, if the previous level was well-tolerated by the patient.
  Arms: BFR-Walking
Other: Conventional therapy — Participants will perform 12 training sessions over 6 weeks. Patients will perform assisted over-ground walking for a total of around 40 minutes, inserted between a 10-minute warm-up and cool-down period. The patient will be encouraged by the same experienced physiotherapist to walk back and forth on 50-meter indoor flat corridor with their habitual walking device. Patient will be asked to walk without stopping until reaching an effort corresponding to a value of 8 out of 10 of the rating of perceived exertion (Borg scale). When the exertion level is reached, the patients will be allowed to rest sitting on a chair if necessary; after a suitable rest period, when patients express sufficient desire to start again, the training will restart
  Arms: Conventional therapy

SUMMARY:
The aim of the study is to evaluate the safety, feasibility and initial efficacy of an interval-based walking training at low speed performed with blood flow restriction (BFR) on gait speed and functional impairments in patients with Multiple Sclerosis (MS).

Patients with severe MS will be recruited at outpatient rehabilitation clinics (University Hospital of Ferrara). Eligible participants will be randomized to interval walking training with BFR (the experimental group) or conventional exercise therapy (the control group) according to a blocked-randomization stratified by gender with 1:1 ratio. Both groups will receive 12 rehabilitative sessions over 6 weeks, for a 2 sessions/week pattern.

The experimental group will undergo interval-based walking training at a slow speed according to a walk:rest ratio of 1:1 for a total of 6 minutes, to be repeated 5 times. Blood flow restriction, applied to the proximal thigh, will be set at a maximum of 40% of systolic blood pressure. The control group will be treated with conventional therapy.

Changes in gait speed, endurance, balance, lower limbs strength and quality of life will be assessed at baseline, at the end of training, and at follow up.

The proposed training modality has never been tested in patients with MS and, if the hypotheses were supported by the results, might be a novel tool to improve muscle strength with a positive impact on gait disabilities, balance and quality of life for patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* primary and secondary progressive MS patients according to the diagnostic MS criteria revised by Polman et al.
* Male and females, aged 18 to 65 years;
* Severe gait impairments, defined by an Expanded Disability Status Scale (EDSS) ranging from 5.5 to 6.5;
* Lack of MS worsening in the previous three months prior to the intervention period;
* Cognitive functioning to provide informed consent identified by a Mini-Mental Status Examination (MMSE) score = 24/30.

Exclusion Criteria:

* Neurologic conditions in addition to MS that may affect motor function and other medical conditions likely to interfere with the ability to complete safely the study protocol, independently from the group assignment;
* Considerable muscle spasticity, defined by a Modified Ashworth Scale (MAS) score > 3 or contractures that may limit range of motion or function for hip, knee or ankle flexors/extensor;
* Relapsing of MS-related conditions or changes in drug therapy or any other confounding factor during the study;
* Rehabilitation treatments or Botulinum toxin injections during the three months preceding the start of the study.
* Intermittent claudication and peripheral artery disease
* Contraindication to exercise training (e.g., unstable angina, congestive heart failure)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Timed 25-foot Walk test | Baseline (prior to the first exercise session, T0); end of the treatment (after 6 weeks, T1); follow-up (after 12 weeks)
  The patient will be directed to one end of a clearly marked 25-foot course and will be instructed to walk 25 feet (7.62 m) as quickly as possible, but safely, using the prescribed assistive devices. The task is immediately administered again by having the patient walk back the same distance. The test will be performed according to the instructions reported on the manual of the National Multiple Sclerosis Society. To ensure an accurate and objective measure of the primary outcome, the time needed for each subject to complete the test will be collected with the aid of a photocells system with a precision of a millisecond and simultaneously by the assessors with a chronometer. The walking speed will be calculated as the mean of the two trials performed.

SECONDARY OUTCOMES:
6-Minute Walking Test | Baseline (prior to the first exercise session, T0); end of the treatment (after 6 weeks, T1); follow-up (after 12 weeks)
  Subjects will be instructed to walk up and down as far as possible on a 22m walkway in six minutes without encouragement, with the possibility to slow down and rest if necessary. The total distance walked will be recorded.
Berg Balance Scale | Baseline (prior to the first exercise session, T0); end of the treatment (after 6 weeks, T1); follow-up (after 12 weeks)
  To evaluate the ability to maintain balance statically or while performing functional movement. It includes 14 observable tasks common to an everyday life measured on a 5-point ordinal scale.
5-time Sit-to-Stand test | Baseline (prior to the first exercise session, T0); end of the treatment (after 6 weeks, T1); follow-up (after 12 weeks)
  Patient stand on a 43-cm chair with his/her arms folded across the chest and the back against the chair. Then the patient will be instructed as follow: "I want you to stand up and sit down 5 times as quickly as you can". The time to complete the 5 repetitions will be recorded.
Multiple Sclerosis Impact Scale | Baseline (prior to the first exercise session, T0); end of the treatment (after 6 weeks, T1); follow-up (after 12 weeks)
  This is a 29-item self-report measure with 20 items associated with a physical function scale and 9 items with a psychological function scale. Items ask about the impact of MS on everyday life in the past two weeks with possible answers set on a 1-5 Likert scale. Each of the two scales is converted to a 0-100 scale where a score of 100 indicates a greater impact of disease on daily function.
Fatigue Severity Scale | Baseline (prior to the first exercise session, T0); end of the treatment (after 6 weeks, T1); follow-up (after 12 weeks)
  The scale consists of answering short questions that require the subject to read each statement and rate his or her level of fatigue from 1 to 7, depending on how appropriate they felt the statement applied to them over the preceding week.
Short Form Health Survey 36 | Baseline (prior to the first exercise session, T0); end of the treatment (after 6 weeks, T1); follow-up (after 12 weeks)
  This is a generic measurement to assess health-related quality of life. It consists of 8 sub-scales with a score ranging from 0-100 used separately as outcome measures of various aspects of health-related-quality of life. It also measures two main health concepts: physical and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Manfredini, MD, Principal Investigator — University Hospital of Ferrara
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published at the end of the trial after deidentification. The database of the study will be published in a public repository.
Supporting Information: SAP
Time Frame: IPD will be available beginning 6 months following study results publication.
Access Criteria: Anyone who wishes to access the data